CLINICAL TRIAL: NCT04400747
Title: The Effects of Single High-dose or Daily Low Dosage Oral Colecalciferol Treatment on Muscle Strength, Muscle Thickness and Independence in Spinal Cord Lesion
Brief Title: Oral Colecalciferol Treatment in Spinal Cord Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Demet Ferahman, Assistant doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMRIST
Record Dates: First submitted 2020-05-17; First posted 2020-05-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injury
Keywords: 25(OH)D; hand grip strength; Spinal cord injuries; muscle thickness
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Sixty patients with spinal cord injury with serum 25 (OH) D3 levels less than 20 ng / ml will be included in the study. One of the treatment groups will receive 6,000 IU of vitamin D daily, and the other group 50000 IU of vitamin D per week for 8 weeks. 20 Patients who don't receive vitamin D will be included in the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- weekly treatment group (Experimental): Twenty patients with spinal cord injury with serum 25 (OH) D3 level less than 20 ng / ml will receive 50,000 IU of vitamin D weekly for 8 weeks.
  Interventions: Drug: Vitamin D3
- daily treatment group (Experimental): Twenty patients with spinal cord injury with serum 25 (OH) D3 level less than 20 ng / ml will receive 6,000 IU of vitamin D daily for 8 weeks.
  Interventions: Drug: Vitamin D3
- control group (No Intervention): 20 patients with high calcium (Ca) values in blood tests, patients with kidney and urinary stones, as well as patients who refuse to use vitamin D supplements will be included in the control group

INTERVENTIONS:
Drug: Vitamin D3 — one group will take weekly oral 50000 IU Vitamin D3, other group will take daily oral 6000 IU Vitamin D3.
  Other Names: cholecalciferol
  Arms: daily treatment group; weekly treatment group

SUMMARY:
Low vitamin D is frequently seen in patients with spinal cord injury (SCI) in acute and chronic periods. Among its causes are insufficient sun exposure, limited oral intake, obesity, the effect of the drugs used on the absorption of vitamin D, kidney and liver diseases. If we consider patients with spinal cord injuries in Turkey, it is difficult to get involved in the society, low exposure to the sun, lack of necessary health controls and immobility brings extra risk factors for the low vitamin D compared to the general population. Despite Turkey Endocrinology and Metabolism Endocrine Society and the International Endocrine Association clinical practice guidelines do not provide specific recommendations about vitamin D, for individuals with spinal cord injuries. Individuals with SCI are at high risk for low vitamin D. Vitamin D levels need to be checked and replaced. Vitamin D doses, application methods and dose intervals used in Physical Therapy and Rehabilitation clinics are different. The aim of our study is to perform the necessary vitamin D replacement for individuals with SCI who have vitamin D deficiency in different dose intervals and to compare the effects of muscle strength, muscle thickness and functional independence with the control group.

DETAILED DESCRIPTION:
Paraplegic patients who admitt to our Physical Therapy and Rehabilitation Clinic, will be included in the rehabilitation program. Sixty spinal cord injured patients with serum 25 (OH) D3 levels less than 20 ng / ml will be included in the study. One of the treatment groups will receive 6,000 IU of vitamin D daily, and the other group 50,000 IU of vitamin D per week for eight weeks. Patients with high calcium (Ca) values in blood tests, patients with kidney stones and urinary stones in urinary ultrasonography (USG) to be performed routinely, as well as patients who refuse to use vitamin D supplements will include in the control group. Spinal cord independence measure (SCIM version 3) will be filled in at the beginning and at the end of 8 weeks to all participants. Jamar Dynamometer will be measured for upper extremity muscle strength, and biceps brachii and triceps muscle thicknesses will be measured by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old
2. Thoracic level chronic spinal cord injury
3. A, B, C, D complete / incomplete patients according to ASIA classification
4. 25 (OH) D3 level in serum is <20 ng / ml
5. Complete muscle strength in upper extremity

Exclusion Criteria:

1. Individuals with chronic liver, kidney, respiratory and parathyroid disease
2. Chronic constipation
3. Patients who have recently used vitamin D
4. Use of drugs that will affect vitamin D and Ca level (Thiazide group diuretics, statins)
5. Acute inflammation (may show false low in vitamin D levels)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 8 weeks
  Measurement of both hands grip strength by Jamar dynamometer

SECONDARY OUTCOMES:
Spinal cord İndependence Measurement (SCIM version 3) | 8 weeks
  The SCIM has been developed to address three specific areas of function in patients with spinal cord injuries (SCI). It looks at self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and a patient's mobility abilities (bed and transfers and indoors/outdoors).
Muscle thickness | 8 weeks
  Both sides biceps brachii and triceps muscle thicknesses will be measured by ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Ferahman, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hummel K, Craven BC, Giangregorio L. Serum 25(OH)D, PTH and correlates of suboptimal 25(OH)D levels in persons with chronic spinal cord injury. Spinal Cord. 2012 Nov;50(11):812-6. doi: 10.1038/sc.2012.67. Epub 2012 Jun 19. PMID 22710945
- [Background] Bauman WA, Zhong YG, Schwartz E. Vitamin D deficiency in veterans with chronic spinal cord injury. Metabolism. 1995 Dec;44(12):1612-6. doi: 10.1016/0026-0495(95)90083-7. PMID 8786732
- [Background] Lamarche J, Mailhot G. Vitamin D and spinal cord injury: should we care? Spinal Cord. 2016 Dec;54(12):1060-1075. doi: 10.1038/sc.2016.131. Epub 2016 Sep 20. PMID 27645263
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Bauman WA, Morrison NG, Spungen AM. Vitamin D replacement therapy in persons with spinal cord injury. J Spinal Cord Med. 2005;28(3):203-7. doi: 10.1080/10790268.2005.11753813. PMID 16048137